CLINICAL TRIAL: NCT00413686
Title: A Phase I Open Label Multi Center Dose Escalation Study to Assess Safety, Tolerability, and Pharmacokinetics of AZD7762 Administered as a Single Intravenous Agent and in Combination With Weekly Standard Dose Gemcitabine in Patients With Advanced Solid Malignancies
Brief Title: Study to Assess Safety of AZD7762 Administered Alone and in Combination With Gemcitabine in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1040C00002
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Solid Tumors
Keywords: Mixed solid tumors
MeSH Terms: interventions — 3-(carbamoylamino)-5-(3-fluorophenyl)-N-(3-piperidyl)thiophene-2-carboxamide; Gemcitabine

ARMS (1):
- 1 (Experimental): AZD7762 monotherapy followed by AZD7762 + gemcitabine
  Interventions: Drug: AZD7762; Drug: Gemcitabine

INTERVENTIONS:
Drug: AZD7762 — intravenous infusion
Drug: Gemcitabine — weekly intravenous infusion
  Other Names: Gemzar®; Gemcitabine HCL

SUMMARY:
This is an open-label, multi-center, dose-escalation, Phase I study to evaluate the safety, tolerability, and pharmacokinetics and to investigate biomarker changes of AZD7762 administered as a single intravenous unit and in combination with gemcitabine. The study is sponsored by AstraZeneca.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* ECOG performance status of 0 or 1
* Patient and tumor type must be suitable for treatment with weekly standard gemcitabine.

Exclusion Criteria:

* Inadequate bone marrow reserve, inadequate liver function or impaired renal function
* Any troponin elevation (above normal range)
* Stage II, III, or IV cardiac status, according to New York Heart Association (NYHA) classification; recent history (ie, within 6 months) of coronary artery disease or arteriosclerotic cardiovascular disease (angina, myocardial infarction [MI])
* Any prior anthracycline treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD7762 alone and in combination with Gemcitabine | Assessed after each course of treatment

SECONDARY OUTCOMES:
To determine the single-dose (after the first single-agent dose) and combination-dose (afer the 2nd combination dose) pharmacokinetics (PK) of AZD7762. | Assessed after each course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, M.D., Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan